CLINICAL TRIAL: NCT05591703
Title: Clinical Outcomes Following Transcutaneous Auricular Neurostimulation to Improve Relapse Prevention: A Long-term Follow-up Study
Acronym: RESTOREb
Status: Completed | Type: Observational
Sponsor: Spark Biomedical, Inc. (Industry)
Collaborators: Hazelden Betty Ford Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: SBM-OWP-03b
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Opioid Use Disorder; Relapse
Keywords: relapse prevention
MeSH Terms: conditions — Opioid-Related Disorders; Recurrence | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants randomized to receive tAN therapy in SBM-OWP-03 Phase II
  Interventions: Behavioral: Clinical Outcomes and Questionnaires
- Participants not randomized to receive tAN therapy in SBM-OWP-03 Phase II
  Interventions: Behavioral: Clinical Outcomes and Questionnaires

INTERVENTIONS:
Behavioral: Clinical Outcomes and Questionnaires — Clinical patient-reported outcomes will be administered remotely at specified timepoints. No treatment or intervention will be administered in this protocol.

SUMMARY:
This is a prospective, observational, longitudinal study to assess clinical outcomes in the 12-months following participants' exit from protocol SBM-OWP-03, Delivering Transcutaneous Auricular Neurostimulation to Improve Relapse Prevention in Opioid Use Disorder (RESTORE; ClinicalTrials.gov Identifier: NCT05053503). Clinical outcome scores will be collected at study exit from protocol SBM-OWP-03, 1 month, 3 months, 6 months, 9 months, and 12 months after study exit from protocol SBM-OWP-03.

ELIGIBILITY:
Inclusion Criteria:

1. Consented participant for protocol SBM-OWP-03, Delivering Transcutaneous Auricular Neurostimulation to Improve Relapse Prevention in Opioid Use Disorder (RESTORE)
2. Participant is English proficient
3. Participant is able to provide informed consent and function at an intellectual level sufficient for study requirements

Exclusion Criteria:

1. Participant is unable to reliably receive and respond to assessments via email or telephone
2. Participant has any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a history of dependence on prescription or non-prescription opioids
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants in Phase II with a relapse event | 12 months (total duration of trial)

SECONDARY OUTCOMES:
Proportion of participants in either Phase I or Phase II with a relapse event | 12 months (total duration of trial)
  Comparison of the proportion of participants in either Phase I or Phase II with a relapse event over the 12-month follow-up period
Mean change in recovery capital measured by Brief Assessment of Recovery Capital (BARC-10) | Baseline to Study Completion (12 months)
  The BARC-10 is a short,10-item measure that examines recovery capital globally. Items were selected from the ARC for the BARC-10 using item response theory. The BARC-10 measures a unidimensional (i.e., global) construct of recovery capital across all the original 10 domains of the ARC. On average, it takes 2-5 minutes to complete. Scores range from 6-60. Individuals who have a recovery capital score of 47 or higher are likely to reach or sustain a year or longer of recovery from substance use disorder.
Mean change in opioid craving measured by the Opioid Craving Scale (OCS) | Baseline to Study Completion (12 months)
  Participants are asked to answer the following three questions with responses ranging from 0-10, where 0=Not at all and 10=Extremely. Total possible score ranges from 0-30 with greater scores indicating higher opioid craving: (1) How much do you currently crave opiates? (2) In the past week, please rate how strong your desire to use opiates has been when something in the environment has reminded you of opiates (example: seeing a medication bottle, using the Internet, visiting a doctor's office, going to a place where you used to buy drugs)? (3) Please imagine yourself in the environment in which you previously used opiates (examples: a party, a hangout, a particular room where you live). If you were in this environment today and if it were the time of day that you typically used opiates, what is the likelihood that you would use opiates today?
Mean change in protracted withdrawal symptoms measured by the Short Opiate Withdrawal Scale-Gossop (SOWS-Gossop) | Baseline to Study Completion (12 months)
  The SOWS-Gossop is an appropriate, precise, and sensitive measure to evaluate the symptoms of acute opioid withdrawal in research or clinical settings. The scale was derived from the original 32-item Opiate Withdrawal Scale to reduce redundancy while providing an equally sensitive measure of opioid withdrawal symptom severity appropriate for research and clinical practice. The assessment is a self-administered test used for the assessment of opiate withdrawal symptoms. The scale contains ten items: yawning, muscular tension, runny eyes, muscle twitching, pains, and aches, feeling of coldness, stomach cramps, insomnia, heart pounding, and feeling sick, making it easy and rapid to administer. The tool has a 4-point rating scale: 0 for 'none,' 1 for 'mild,' 2 for 'moderate,' and 3 for 'severe', with scores ranging from 0 to 30.
Mean change in depression symptoms across time measured by Patient Health Questionnaire (PHQ-9) | Baseline to Study Completion (12 months)
  The PHQ-9 is a validated tool in mental health and considered a powerful tool to assist clinicians with diagnosing depression and monitoring treatment response. The relationship between opioid use and depression is bidirectional. The PHQ-9 is a nine-item depression scale and is based directly on the nine diagnostic criteria for major depressive disorder in the DSM-IV. Each of the nine items is rated on a 0 (not at all) to 3 (nearly every day) scale. A total score is calculated by summing the nine items. Scores range from 0 to 27 and higher scores indicate a higher degree of depression.
Mean change in anxiety across time measured by Generalized Anxiety Disorder (GAD-7) | Baseline to Study Completion (12 months)
  The GAD-7 is a valid and efficient tool for screening for GAD and assessing its severity in clinical practice and research. The questionnaire consists of 7 questions in which participants are asked to rate each item on a 0 (not at all) to 3 (nearly every day). GAD-7 total score for the seven items ranges from 0 to 21 where 0-4 represents minimal anxiety, 5-9 represents mild anxiety, 10-14 represents moderate anxiety and 15-21 represent severe anxiety.
Mean change in PTSD symptoms across time measured by the PTSD Checklist for DSM-5 (PCL-5) | Baseline to Study Completion (12 months)
  Symptoms of post-traumatic stress disorder (PTSD) and opiate dependency may overlap, to which, opioid withdrawal symptoms may emulate PTSD hyperactive startle response. This is indicative a common physiological mechanism. The PCL-5 scale is the gold standard in PTSD assessment. It consisted of a 20-item self-report measurement that is capable of measuring symptom change during and after treatment. Additionally, the scale can provide a provisional PTSD diagnosis. Each of the 20 items is rated on a 0 (not at all) to 4 (extremely) scale. A total symptom severity score is calculated by summing the 20 items. Scores range from 0 and 80 and higher scores indicating a higher degree of PTSD symptomology. Evidence suggests that a10 to 20-point reduction in score represents a clinically significant change in PTSD symptoms.
Mean change in Quality of Life across time measured by World Health Organization Quality of Life(WHOQOL-BREF) domain scores | Baseline to Study Completion (12 months)
  The WHOQOL-BREF is a shorter version of the original assessment tool and is commonly used in clinical trials with participants undergoing substance use disorder intervention. The WHOQOL-BREF is comprised of 26-items and assesses the participant's quality of life across specific domains: physical health, psychological health, social relationships, and environment.24 In addition, there are 2 items that measure overall quality of life and general health. Participants rate how much they have experienced each item in the preceding two weeks on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely). Domain scores are scaled in a positive direction with higher scores denoting higher quality of life. The mean score of items within each domain is used to calculate the domain score. Raw domain scores will be converted to a 0 to 100 scale.
Mean change in Commitment to Sobriety Scale (CSS-5) | Baseline to Study Completion (12 months)
  Ratings of participant-perceived level of motivation and dedication to achieving initial and maintaining on-going sobriety for substance use will be measured using the 5-item Commitment to Sobriety Scale (CSS-5). Each statement is rated on a 6-point Likert scale, ranging from 1 (strongly disagree) to 6 (strongly agree). Example items include: "Staying sober is the most important thing in my life" and "I will do whatever it takes to recover from my addiction." Following the completion of the CSS-5, participants will be asked to reflect and rate level of confidence on their commitment to abstinence for the next 30 days using a 10-point scale, from 1 (not at all confident) to 10, (very confident).

OTHER OUTCOMES:
Record traumatic life events measured by the Life Events Checklist for DSM-5 (LEC-5) | Baseline to Study Completion (12 months)
  The Life Events Checklist for DSM-5 (LEC-5) is a self-report measure designed to screen for potentially traumatic events in a respondent's lifetime. The LEC-5 assesses exposure to 16 events known to potentially result in PTSD or distress and includes one additional item assessing any other extraordinarily stressful event not captured in the first 16 items.
Record self-report of peer recovery support engagement | Baseline to Study Completion (12 months)
  Participants will be asked about their engagement in peer recovery support groups through one-item: "How often have you attended peer recovery support groups or services (examples include, formal peer recovery support services, 12-step meetings, faith-based recovery support, SMART recovery, and other mutual-aid groups engagement) since your last survey date?" Participants will be given a 6-point ordinal response scale: Daily, Four or more times per week, One to three times per week, Two to four times per month, Once a month or less, or Never.
Record self-report of MOUD prevalence and adherence | Baseline to Study Completion (12 months)
  Participants will be asked if they are currently receiving MOUD treatment. For those that are, follow up questions will ask participants to report on type and kind of medication they are taking, as well as their current adherence and rationale for any reported deterrence from physician-prescribed treatment. "Do you have a prescription for an anti-craving medication?"; "Which of the following medications are you currently prescribed?". Example items related to adherence: "Have you been able to take your medication as prescribed?", "Which of the following medications have you NOT taken as prescribed?", and "What is the reason that you have not taken your anti-craving medication as prescribed?" For adherence rationale, respondents are given five response options, including an Other category in which they can provide a short answer option unique to their situation.
Proportion of participants who qualify for a change in ICD-10 code | Baseline to Study Completion (12 months)
  Responses to the above questionnaires will be reviewed against the DSM-5 and ICD-10 code definitions. If a participant qualified for a change in ICD-10 code, the original and projected ICD-10 code changes will be recorded.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Betty Ford Foundation, Rancho Mirage, California
  - Hazelden Betty Ford Foundation, Center City, Minnesota
  - Hazelden Betty Ford Foundation, Plymouth, Minnesota

IPD SHARING:
Plan to Share IPD: No